CLINICAL TRIAL: NCT07225335
Title: Impact of OptiCreatine on Plasma Creatine and Gastrointestinal Effects in Males and Females
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TSI Group LTD (Industry)
Collaborators: University of North Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 25-2972
Record Dates: First submitted 2025-11-03; First posted 2025-11-06 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Creatine Absorption in Healthy Adults
Keywords: Absorption; creatine; Healthy adults
MeSH Terms: interventions — Creatine

STUDY DESIGN:
Intervention Model Description: Acute: In a randomized double-blind, cross-over design, participants will be randomly assigned using a using a computer-generated randomization scheme to consume either OptiCreatine or creatine monohydrate supplement. All participants will complete both treatments, including a minimum of a 3-day washout period.
  Chronic: In a randomized double-blind design, participants will be randomly assigned using block randomization in a 1:1 fashion to participants in a creatine loading dose of OptiCreatine or creatine monohydrate.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OptiCreatine (Experimental): Combines creatine with other bioactive compounds purported to enhance absorption.
  Interventions: Dietary Supplement: OptiCreatine
- Creatine monohydrate (Active Comparator)
  Interventions: Dietary Supplement: Creatine Monohydrate

INTERVENTIONS:
Dietary Supplement: OptiCreatine — OptiCreatine is a formulation, which combines creatine with other bioactive compounds purported to enhance absorption.
  Arms: OptiCreatine
Dietary Supplement: Creatine Monohydrate — Creatine monohydrate (Creapure®)
  Arms: Creatine monohydrate

SUMMARY:
The study aims to evaluate the novel OptiCreatine formulation, which combines creatine with other bioactive compounds purported to enhance absorption and reduce gastrointestinal (GI) discomfort. Using a randomized, double-blind, crossover design, the study will compare the acute and chronic effects of OptiCreatine versus Creatine monohydrate in healthy, recreationally active adults. Participants will be asked to orally consume both the OptiCreatine and the creatine monohydrate. Primary outcomes include plasma creatine concentrations, gastrointestinal symptomatology, and fluid distribution measured through bioelectrical impedance spectroscopy.

DETAILED DESCRIPTION:
The study aims to evaluate the novel OptiCreatine formulation, which combines creatine with other bioactive compounds purported to enhance absorption and reduce gastrointestinal (GI) discomfort. The study objectives are as follows:

* Aim 1: To examine the acute effects of OptiCreatine compared to creatine monohydrate on plasma creatine concentrations and gastrointestinal symptoms.
* Aim 2: To example the effects of 5-days of creatine loading with OptiCreatine compared to creatine monohydrate on gastrointestinal symptoms and fluid distribution.

General Design: All data collection will be completed by the Principal Investigator and Research Assistants at the University of North Carolina. Participants will be asked to report to the Applied Physiology Laboratory and Human Performance Center for enrollment and testing sessions. Thirty-two individuals total will be enrolled into the study. Sixteen participants will be enrolled into the acute phase; Sixteen will be enrolled into the chronic phase with random assignment to OptiCreatine (n=8) or creatine monohydrate (n=8). Participants from the acute phase are eligible to enroll into the chronic phase. The acute phase will require 2 in person visits, in random order, with participants randomly assigned in a cross-over fashion to OptiCreatine vs creatine monohydrate. Blood samples will be obtained at baseline and at 0.5, 1, 1.5, 2, 3, 4, and 5 hrs. following ingestion of the assigned treatment. A minimum of 72 hrs. will take place in between acute visits. For the chronic phase, participants will complete baseline assessments for GI symptoms via questionnaires (bloating questionnaire, gastrointestinal symptom rating scale, digestion associated quality of life questionnaire) and fluid distribution from multi-frequency bioelectrical impedance analysis (MF-BIA). Following baseline testing, participants will be randomly assigned to an OptiCreatine or creatine monohydrate group. Post testing evaluation will occur within 48 hours of the 5-day loading phase.

Supplementation Phase:

* Acute: In a randomized double-blind, cross-over design study, participants will be randomly assigned using a using a computer-generated randomization scheme to consume either OptiCreatine (5 g + 6 oz water, n=8) or creatine monohydrate supplement (5 g + 6 oz water, n=8). All participants will complete both treatments, including a minimum of a 3-day washout period.
* Chronic: In a randomized double-blind design study, participants will be randomly assigned using block randomization in a 1:1 fashion using a computer generation randomization scheme to participants in a creatine loading dose (4 x 5 grams daily- 20 g per day for 5 days) of OptiCreatine or creatine monohydrate.

Participants will be asked to arrive at the laboratory for all visits after a minimum 8-hour fast from caloric foods and beverages, 48-hour abstention from vigorous exercise, and 24-hour abstention from caffeine consumption. Participants will be asked to maintain normal dietary intake along with no more than 200mg of caffeine per day for the duration of the study. Measurements of anthropometrics, GI symptoms, and fluid distribution will be obtained. For the acute phase, blood samples will be taken from the antecubital region.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 18-45 yrs
* Body mass index of <35 kg/m2
* Recreationally active [≥30 minutes of moderate-intensity physical activity per week as defined by the International Physical Activity Questionnaire (IPAQ)]
* Participant is healthy and free from disease as determined by a health history questionnaire.
* Participant agrees to abstain from caffeine (24 hrs. prior), tobacco (24 hrs. prior), and alcohol (24 hrs. prior) before testing days

Exclusion Criteria:

* Has chronic kidney disease, liver disease, chronic obstructive pulmonary disease, or cancer
* Currently using medications that may directly impact the primary outcomes including: diuretics and corticosteroids)
* Currently using creatine monohydrate
* Has severely impaired hearing or speech or inability to speak English

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-11-07 (Estimated); Primary Completion 2026-05-10 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic Outcomes: Concentration maximum (Cmax) | Over a period of 5 hrs. post dose of creatine
  the maximum observed plasma concentration (Cmax)
Pharmacokinetic Outcomes: Time to concentration maximum (Tmax) | Over a period of 5 hrs. post dose of creatine
  The time to reach the maximum observed plasma concentration
Pharmacokinetic Outcomes: Area Under the Curve (AUC) | Over a period of 5 hrs. post dose of creatine
  The area under the concentration-time curve (AUC)

SECONDARY OUTCOMES:
Digestion-associated Quality of Life Questionnaire (DQLQ) assessment | 6 days
  Digestion-associated Quality of Life Questionnaire (DQLQ) will be assessed on a scale of 0% to 100% at baseline and 6 days, with 0% indicating no effect (never) on digestion-associated quality of life to 90%-100% (always effecting digestion-associated Quality of Life)
Self-perception questionnaire for assessment of bloating | 6 days
  Assessment of bloating using a self-perception questionnaire on a scale of None (no bloating) to very severe (severe bloating) will be conducted at the 1st study visit (baseline), at the 2nd study visit (6 days) after 5 days of creatine loading.
Gastrointestinal Symptom Rating Scale (GSRS) | 6 days
  Gastrointestinal Symptom Rating Scale (GSRS) will be conducted at the 1st study visit (baseline), at the 2nd study visit (6 days) after 5 days of creatine loading. The GSRS is a disease-specific instrument of 15 items combined into five symptom clusters depicting Reflux, Abdominal pain, Indigestion, Diarrhea and Constipation. The GSRS has a seven-point graded Likert-type scale where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms.

OTHER OUTCOMES:
Fluid distribution, Total Body water | Baseline and after 6 days
  A multi-frequency bioelectrical impedance spectroscopy (BIA) device will be used (InBody770) to measure fluid distribution. Device software will automatically estimate total body water (TBW), intracellular fluid (ICF), and extracellular fluid (ECF). The fluid distribution will be expressed in liters (L)
Height | Baseline at day 6
  The height of the participants will be measured for the determination of BMI, kg/m2. Height will be measured in meters (m).
Weight | Baseline and Day 6
  The weight of the participants will be measured for the determination of BMI, kg/m2. Weight will be measured in kilograms (m). Weight will also be used in the body water distribution calculations.
Fluid distribution, Intracellular fluid | Baseline and after 6 days
  A multi-frequency bioelectrical impedance spectroscopy (BIA) device will be used (InBody770) to measure fluid distribution. Device software will automatically estimate total body water (TBW), intracellular fluid (ICF), and extracellular fluid (ECF). Water distribution will be expressed in liters (L).
Fluid distribution, Extracellular fluid | Baseline and 6 days
  A multi-frequency bioelectrical impedance spectroscopy (BIA) device will be used (InBody770) to measure fluid distribution. Device software will automatically estimate total body water (TBW), intracellular fluid (ICF), and extracellular fluid (ECF). Water distribution will be expressed in liters (L).

CONTACTS AND LOCATIONS:
Overall Officials: John A Rathmacher, Ph.D., Study Director — TSI Group LTD
Locations (1):
- Applied Physiology Laboratory (Fetzer Hall, Room 025), Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No